CLINICAL TRIAL: NCT07364669
Title: A Randomized, Double-Blind, Cross Over Study to Assess Pharmacokinetic and Pharmacodynamic Effects of Insulex® R in Comparison to Humulin® R in Healthy Subjects
Brief Title: Pharmacokinetic and Pharmacodynamic Effects of Insulex® R in Comparison to Humulin® R in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Pisa S.A. de C.V. (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PROT/01-INSR-24/01
Record Dates: First submitted 2025-12-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects
Keywords: Recombinant Human Insulin; Bioequivalence; Euglycemic Clamp; Pharmacokinetics (PK); Pharmacodynamics (PD); Short-Acting Insulin
MeSH Terms: interventions — Biosimilar Pharmaceuticals

STUDY DESIGN:
Intervention Model Description: PK/PD euglycemic glucose clamp
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulex® R (Experimental): Soluble human insulin, biosimilar, 100 IU/mL, single subcutaneous injection of 0.3 IU/kg body weight
  Interventions: Drug: Insulex® R (soluble human insulin, biosimilar)
- Humulin® R (Active Comparator): Soluble human insulin, biosimilar, 100 IU/mL, single subcutaneous injection of 0.3 IU/kg body weight
  Interventions: Drug: Humulin® R (soluble human insulin, biosimilar)

INTERVENTIONS:
Drug: Insulex® R (soluble human insulin, biosimilar) — Investigational insulin, Insulex® R (soluble human insulin, biosimilar)
  Arms: Insulex® R
Drug: Humulin® R (soluble human insulin, biosimilar) — Marketed reference insulin, Humulin® R (soluble human insulin, biosimilar)
  Arms: Humulin® R

SUMMARY:
The goal of this clinical trial is to evaluate whether Insulex® R demonstrates similar pharmacokinetic (PK) and pharmacodynamic (PD) profiles compared to Humulin® R after a single subcutaneous dose of 0.3 units/kg in healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1, randomized, double-blind, two-period, two-sequence crossover clinical trial aims to evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) bioequivalence of Insulex® R compared to Humulin® R after a single subcutaneous dose of 0.3 units/kg in healthy adult subjects. The study was designed in accordance with international regulatory guidelines, including the U.S. Food and Drug Administration (FDA) guidance for demonstrating biosimilarity of insulin products and the European Medicines Agency (EMA) guidelines for the clinical development of biosimilar insulins. Each subject underwent a Screening Visit (Visit 1), two 1-day in-house Treatment Periods (Visit 2 and Visit 3), and a Follow-up Visit (Visit 4) to performed safety procedures. The washout period between Treatment Periods was 7 to 14 days. During each Treatment Period, subjects will receive a single subcutaneous dose of either Insulex® R or Humulin® R under euglycemic glucose clamp conditions. Blood samples will be collected at prespecified intervals to measure serum insulin and C-peptide concentrations. Glucose infusion rates will be monitored continuously to assess PD response. The rigorous assessment of PK and PD profiles under controlled clamp conditions is essential to confirm biosimilarity and ensure therapeutic equivalence. Successful demonstration of bioequivalence will provide a safe, effective, and cost-accessible recombinant human rapid-acting insulin option for patients requiring insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male adults, ages ≥ 18 and ≤ 55 years
2. Body mass index (BMI) ≥ 18.5 kg/m2 to ≤ 27.0 kg/m2 and stable body weight by history for ≥ 3 months (defined as change < 5%)
3. Fasting plasma glucose < 100 mg/dL and HbA1c < 5.7% (based on American Diabetes Association [ADA] criteria; American Diabetes Association, 2023)
4. Female subjects of childbearing potential (WOCBP) must use highly effective contraception as defined in section 9.1.9 Contraception. For surgically sterile subjects (e.g., those who have undergone bilateral tubal ligation, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), the site will attempt to retrieve medical records that document the sterility; however, the absence of records will not exclude the participant. If medical records cannot be obtained, serum and urine pregnancy tests will be performed. For postmenopausal females (no menses > 12 months), postmenopausal status will be confirmed through testing for FSH levels in the menopausal range (as specified by the responsible laboratory) for amenorrheic subjects.
5. Subjects must be able to provide written informed consent and are willing to follow study procedures and commitment to the study duration.

Exclusion Criteria:

1. Pregnant, lactating or intending to become pregnant during the study.
2. Subjects with confirmed diabetes type 1 or type 2.
3. Presence of any clinically significant co-morbidities, or physical exam, ECG, or laboratory findings at screening or upon clinic admission that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of the study results.
4. Active or untreated malignancy or has been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for < 5 years.
5. Supine heart rate > 100 or < 40 beats per minute at screening, based on the average of 3 consecutive measurements.
6. Supine systolic blood pressure > 140 mm Hg or < 90 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg at Screening or upon clinic admission. If blood pressure is outside of the specified ranges, it may be repeated once 20-30 minutes later the same day.
7. Subjects with a prior history of any serious adverse reaction, hypersensitivity to study drugs or drug components.
8. History of any major surgery within 6 months prior to screening, per Investigator discretion.
9. History of any active infection, other than mild viral illness within 30 days prior to the first dose of study drug as judged by the Investigator.
10. History of any active infection, other than mild viral illness within 30 days prior to the first dose of study drug as judged by the Investigator.
11. History of regular use of nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipe, chewing tobacco, nicotine patch or gum) or vaping products within 3 months prior to check-in for the first in-house period. Subjects must refrain from using nicotine-containing products until after the completion of the Follow-Up Visit after the last dose of study drug.
12. History of drug abuse as judged by the Investigator or a positive urine drug test at Screening or upon clinic admission. Frequent use of marijuana or other tetrahydrocannabinol (THC) products within 6 weeks, or clinically under the effect at screening or upon clinic admission, as per Investigator evaluation or a positive urine drug test at Screening or upon clinic admission.
13. History of or positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2) antibody.
14. Subject is not able to avoid physical activity, avoid alcohol, caffeinated drinks, smoking or medication other than the study medication for 24 hours prior to and throughout the treatment period. (Herbal products and non-routine vitamins are not allowed within 14 days prior to dosing. Routine vitamins are permitted up to 48 hours prior to dosing. Chronic use of acetaminophen is excluded, but occasional use is permitted.) Adequate washout for any concomitant medication that may impact insulin's effect on blood glucose must be ensured and such medications cannot be used throughout the treatment period.
15. Laboratory or clinical evidence of current infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), i.e., COVID-19, at Screening or upon clinic admission or administration of an approved, authorized, or emergency use approved COVID-19 vaccine within 14 days prior to dosing with study drug.
16. Any anticipated/planned procedures (e.g., surgery), that interfere with the compliance or the subject's ability to complete the study.
17. Participation in an investigational study within 30 days prior to dosing or 5 half-lives within the last dose of investigational product whichever is longer.
18. Have previously participated, completed, or withdrawn from this study.
19. Donation or loss of > 500 mL of whole blood within 8 weeks, platelets within 2 weeks and plasma within 4 weeks of the first dose of study drug. Receipt of blood products within 2 months prior to check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
AUCINS_0-12h | 12 hours
  Area under the insulin concentration - time curve (AUC) from 0 to 12 hours; primary endpoint to assess PK profile according EMA guideline
Cmax | 12 hours
  Maximum insulin concentration; primary endpoint to assess the PK profile according EMA guideline
AUCGIR_0-12h | 12 hours
  Area under the glucose infusion rate (GIR) time curve from 0 to 12 hours; primary endpoint to assess the PD profile according EMA guideline
GIRmax | 12 hours
  Maximum Glucose Infusion Rate; primary endpoint to assess PD profile according EMA guideline

SECONDARY OUTCOMES:
AUCINS_0-2h | 4 hours
  Area under the partial insulin concentration - time curves (AUC) from 0 to 4 hours; to assess PK profile
AUCINS_0-6h | 6 hours
  Area under the partial insulin concentration - time curves (AUC) from 0 to 6 hours, to assess PK profile
AUCINS_6-12h | 6 hours
  Area under the partial insulin concentration - time curves (AUC) from 6 to 12 hours; to assess PK profile
AUCINS_0-∞ | 12 hours
  Area under the serum insulin concentration curve from 0 to infinity (if possible); to assess PK profile
Tmax | 12 hours
  Time to maximum insulin concentration; to assess PK profile
t50%-INS (early) | 12 hours
  Time to half-maximum insulin concentration before maximum insulin concentration (Cmax); to assess PK profile
t50%-INS (late) | 12 hours
  Time to half-maximum insulin concentration after maximum insulin concentration(Cmax); to assess PK profile
t½ | 12 hours
  Terminal elimination half - life; to assess PK profile
λz | 12 hours
  Terminal elimination rate constant; to assess PK profile
AUCGIR_0-2h | 2 hours
  Area under glucose infusion rate (GIR) time curve from 0 to 2 hours; to assess PD profile
AUCGIR_0-6h | 6 hours
  Area under glucose infusion rate (GIR) time curve from 0 to 6 hours; to assess PD profile
AUCGIR_6-12h | 6 hours
  Area under glucose infusion rate (GIR) time curve from 6 to 12 hours; to assess PD profile
tGIR_max | 12 hours
  Time to maximum glucose infusion rate (GIR); to assess PD profile
t50%-GIR (early) | 12 hours
  Time to half - maximum glucose infusion rate (GIR) before maximum glucose infusion rate (GIRmax); to assess PD profile
t50%-GIR (late) | 12 hours
  Time to half - maximum glucose infusion rate (GIR) after maximum glucose infusion rate (GIRmax); to assess PD profile
tGIR_onset | 12 hours
  Time to start of glucose infusion rate (GIR) post - dose; to assess PD profile
Adverse Events | From screening to follow-up visit (up to 30 days after Visit 1)
  The number and percentage of subjects with TEAEs will be summarized by MedDRA-coded SOCs and PTs. All TEAEs will be assessed for severity and for relation to study drug.
Number of participants with clinical findings on physical examination from baseline (screening) to follow-up visit. | From screening to follow-up visit (up to 30 days after Visit 1)
  Physical examination findings considered clinically significant by the PI will be summarized by body system with counts and percentages of subjects for values at treatment visits.
Number of participants with significant changes observed from baseline (screening) to follow-up visit in safety laboratory results (hematology, biochemistry, and urinalysis) for each analite. | From screening to follow-up visit (up to 30 days after Visit 1)
  Value outside the normal range (as defined by the laboratory) or deemed clinically significant at the Investigator's discretion in safety laboratory results (hematology, serum chemistry, urinalysis) will be recorded and reported as the number of participants with significant changes in safety laboratoriy results.
Number of participants with significant changes observed from baseline (screening) to follow-up visit in ECG parameters. | From screening to follow-up visit (up to 30 days after Visit 1)
  The following parameters will be recorded from thsubject's ECG trace as calculated by the machine algorithm: heart rate, QT interval, PR interval, QRS interval, RR interval, and QTc (corrected) using the Fridericia correction.
Injection site reactions | From screening to follow-up visit (up to 30 days after Visit 1)
  Evaluated quantitatively using the Grading Scale for Injection Site Reaction (based on the Guidance for Industry-Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, 2007); which assesses pain, tenderness, erythema/redness, and swelling on a four-point scale: Grade 1 - Mild (does not interfere with activity), Grade 2 - Moderate (interferes with activity/discomfort when moving), Grade 3 - Severe (significant discomfort at rest), and Grade 4 - Potentially Life Threatening (Emergency Room visit or hospitalization). For erythema and swelling, the local reaction measured at the single largest diameter should be recorded.
  .
Number of participants with significant changes observed from baseline (screening) to follow-up visit in body temperature. | From screening to follow-up visit (up to 30 days after Visit 1)
  Body temperature in °C. Any clinically significant findings at the investigator's discretion and/or outside the range identified for the vital sign assessment.
Number of participants with significant changes observed from baseline (screening) to follow-up visit in blood pressure. | From screening to follow-up visit (up to 30 days after Visit 1)
  Given by the measurement of systolic and diastolic blood pressure in mmHg. Any clinically significant findings at the investigator's discretion and/or outside the range identified for the vital sign assessment.
Number of participants with significant changes observed from baseline (screening) to follow-up visit in heart rate. | From screening to follow-up visit (up to 30 days after Visit 1).
  Reading taken in beats per minute (bpm) obtained from the oximeter placed on the tip of the index finger. Any clinically significant findings at the investigator's discretion and/or outside the range identified for the vital sign assessment.
Number of participants with significant changes observed from baseline (screening) to follow-up visit in respiratory rate. | From screening to follow-up visit (up to 30 days after Visit 1).
  Reading taken in breaths per minute (bpm) obtained from the oximeter placed on the tip of the index finger. Any clinically significant findings at the investigator's discretion and/or outside the range identified for the vital sign assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Prosciento, Inc, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeWitt DE, Hirsch IB. Outpatient insulin therapy in type 1 and type 2 diabetes mellitus: scientific review. JAMA. 2003 May 7;289(17):2254-64. doi: 10.1001/jama.289.17.2254. PMID 12734137
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Chance RE, Frank BH. Research, development, production, and safety of biosynthetic human insulin. Diabetes Care. 1993 Dec;16 Suppl 3:133-42. doi: 10.2337/diacare.16.3.133. PMID 8299470
- [Result] Vocelka CR, Burdge EC, Kunzelman KS, Thomas R, Verrier ED. An in vitro protocol for evaluation and comparison of membrane oxygenators. J Extra Corpor Technol. 1993;25(4):161-6. PMID 10146588
- [Result] Yamada N, Chung YS, Takatsuka S, Arimoto Y, Sawada T, Dohi T, Sowa M. Increased sialyl Lewis A expression and fucosyltransferase activity with acquisition of a high metastatic capacity in a colon cancer cell line. Br J Cancer. 1997;76(5):582-7. doi: 10.1038/bjc.1997.429. PMID 9303355
- [Result] Colombo TJ, Saward EW, Greenlick MR. The integration of an OEO health program into a prepaid comprehensive group practice plan. Am J Public Health Nations Health. 1969 Apr;59(4):641-50. doi: 10.2105/ajph.59.4.641. No abstract available. PMID 5813452
- [Result] Guerci B, Sauvanet JP. Subcutaneous insulin: pharmacokinetic variability and glycemic variability. Diabetes Metab. 2005 Sep;31(4 Pt 2):4S7-4S24. doi: 10.1016/s1262-3636(05)88263-1. PMID 16389894